CLINICAL TRIAL: NCT02636270
Title: Treatment With Recombinant Human Insulin-like Growth Factor 1 (rhIGF-1) in Patients With Pappalysin-2 (PAPP-A2) Gene Mutation.
Brief Title: IGF-1 Treatment for Individuals With Short Stature Due to PAPP-A2 Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-6218
Record Dates: First submitted 2015-11-10; First posted 2015-12-21 (Estimated); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Short Stature
MeSH Terms: conditions — Dwarfism | interventions — mecasermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PAPP-A2 deficient patients (Experimental): Patients deficient in PAPP-A2 with short stature will be treated with Increlex (rhIGF-1)
  Interventions: Drug: Increlex

INTERVENTIONS:
Drug: Increlex — Treat PAPP-A2 deficient patients with Increlex
  Other Names: rhIGF-1

SUMMARY:
With this study we want to investigate the pharmacokinetic (PK) effect of a single injection of rhIGF-1 in patients with PAPP-A2 mutations compared to heterozygous carriers and healthy controls. This will be followed by treatment of PAPP-A2 deficient patients with IGF-1 for a period of one-year to assess growth velocity. Additionally, we want to further describe the phenotypic characteristics of patients with PAPP-A2 deficiency.

DETAILED DESCRIPTION:
The 24-hour pharmacokinetic response of free and total IGF-1 and IGF binding protein-3 (IGFBP-3) to a single dose of rhIGF-1 (120 mcg/kg) in three patients with PAPP-A2 mutation compared to up to four unaffected heterozygous relatives and 2 healthy adult controls.

One-year trial of rhIGF-1 at standard dose given to the two youngest males with PAPP-A2 mutation. The primary end point of this trial will be first year height velocity. Secondary outcomes will include height standard deviation score (SDS), height velocity, and whole body and lumbar spine bone mineral density assessment. The study was amended to extend the treatment period to continue until the subject has stopped growing (or elects to withdraw). All study procedures remain the same. Important note: the treatment phase continues to follow the youngest affected male. The older affected male developed an adverse event that resulted in discontinuation of treatment.

A post-treatment follow up visit (either in-person or remote) will be completed for the study participant who remained on Increlex approximately one-year after their discontinuation of therapy.

Description of additional phenotypic characteristics of patients with PAPP-A2 mutation will be studied by collecting information on glucose and insulin metabolism, body composition, bone geometry and bone density before and after treatment with rhIGF-1. These measures will be collected at the 12-month time period, and every year thereafter until the completion of the study. All three affected siblings will take part in the phenotyping activities.

ELIGIBILITY:
PAPP-A2 deficient

Inclusion Criteria:

* Defect in PAPP-A2 (heterozygous or homozygous mutation)

Exclusion Criteria:

* None

Healthy Volunteers

Inclusion Criteria:

* Between the ages of 18 and 30
* In general good health

Exclusion Criteria:

* Any medications (with the exception of contraceptives)
* Pregnancy

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Backeljauw, MD, Principal Investigator — Cincinnati Childrens Hospital; Gajanathan Muthuvel, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center

IPD SHARING:
Plan to Share IPD: Yes
De-identifiable data may be shared with physician that is treating the only other two patients in the world with this genetic mutation.
Supporting Information: CSR
Time Frame: The participant data will be available when the treatment trial is actively ongoing. Per study protocol, the study will provide clinical updates to the participants primary Endocrinologist. Should the family request any further information be shared once the study is closed, it can be given to a physician specified by the family.
Access Criteria: De-identifiable data may be shared with physician that is treating the only other two patients in the world with this genetic mutation.

REFERENCES:
- [Result] Muthuvel G, Dauber A, Alexandrou E, Tyzinski L, Andrew M, Hwa V, Backeljauw P. Five-Year Therapy with Recombinant Human Insulin-Like Growth Factor-1 in a Patient with PAPP-A2 Deficiency. Horm Res Paediatr. 2023;96(5):449-457. doi: 10.1159/000529071. Epub 2023 Jan 16. PMID 36646053
- [Result] Cabrera-Salcedo C, Mizuno T, Tyzinski L, Andrew M, Vinks AA, Frystyk J, Wasserman H, Gordon CM, Hwa V, Backeljauw P, Dauber A. Pharmacokinetics of IGF-1 in PAPP-A2-Deficient Patients, Growth Response, and Effects on Glucose and Bone Density. J Clin Endocrinol Metab. 2017 Dec 1;102(12):4568-4577. doi: 10.1210/jc.2017-01411. PMID 29029190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an n=7 study. A total of seven individuals will be recruited to participate in this study. Among the participants, we will have the three affected siblings with Pappalysin-2 (PAPP-A2) mutation (two males and one female), their heterozygous relatives (2 parents) and 2 healthy adult controls.
Pre-assignment Details: Not applicable to this research study. All participants that were eligible for the study and agreed to participate were enrolled.
Groups:
- PAPP-A2 Deficient Patients: Patients deficient in PAPP-A2 will participate in the 24-hour pharmacokinetic study, and those who have not completed growth will be treated with Increlex (recombinant human IGF-1).
- Healthy Control Participants: Healthy controls between the ages of 18-30 will be included in the 24-hour pharmacokinetic study.
- PAPP-A2 Heterozygous Relatives: Unaffected heterozygous PAPP-A2 deficient relatives will be included in the 24-hour pharmacokinetic study.
Period: Overall Study
Arm/Group | PAPP-A2 Deficient Patients | Healthy Control Participants | PAPP-A2 Heterozygous Relatives
Started | 3 | 2 | 2
Completed | 1 | 2 | 2
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — subject had completed growth prior to enrollment, so never started on recombinant IGF-1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PAPP-A2 Deficient Patients: Three siblings with PAPP-A2 deficiency due to homozygous PAPP-A2 mutation. The two younger siblings were recruited for extension trial treatment with recombinant human Insulin-like Growth Factor 1 (IGF-1).
- PAPP-A2 Heterozygous Relatives: Unaffected heterozygous PAPP-A2 deficient relatives (2 parents).
- Health Control Participants: Healthy adult controls with no known variants in PAPP-A2.
- Total: Total of all reporting groups
Arm/Group | PAPP-A2 Deficient Patients | PAPP-A2 Heterozygous Relatives | Health Control Participants | Total
Number analyzed (Participants) | 3 | 2 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 0 | 2
  Between 18 and 65 years | 1 | 2 | 2 | 5
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 2 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 1 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity
Description: Height velocity in a patient with PAPP-A2 deficiency treated with rhIGF-1 for five years (when the patient elected to discontinue treatment after reviewing growth velocity and skeletal maturation). Ultimately only one patient was treated for the study duration with results reported, as the other recruited participant (sibling of the treated patient) experienced pseudotumor cerebri and discontinued treatment after 51 days. He nevertheless was followed, with height velocity also reported.
Time Frame: Yearly until participant on treatment stops growing, or discontinues treatment (up to 6 years)
Population: The untreated comparison sibling was not evaluated at year 5 past completion of growth.
Measure: Number; unit: cm/y
Groups:
- Treatment With rhIGF-1: Patient deficient in PAPP-A2 with short stature treated with recombinant human IGF-1 (rhIGF-1)
- Untreated Comparison: Patient deficient in PAPP-A2 with short stature who was not treated with rhIGF-1 due to development of pseudotumor cerebri (sibling of treated patient)
Arm/Group | Treatment With rhIGF-1 | Untreated Comparison
Number analyzed (Participants) | 1 | 1
cm/y
  Baseline | 3.0 | 4.3
  Year 1 | 6.2 | 4.8
  Year 2 | 5.0 | 5.3
  Year 3 | 5.3 | 3.4
  Year 4 | 7.6 | 1.4
  Year 5: number analyzed (Participants) | 1 | 0
  Year 5 | 6.5 |

2. Secondary Outcome: Height Standard Deviation Score
Description: Height Standard Deviation Score is the standard deviation above or below the mean the height is for age and gender. Values were obtained by plotting heights on Centers for Disease Control and Prevention growth charts. An increase in Height Standard Deviation Score correlates with increase in height. Results are reported for the participant with PAPP-A2 deficiency treated with rhIGF-1, as well as sibling who did not continue treatment with rhIGF-1.
Time Frame: Annually until completion of study, up to 6 years
Population: The participant treated with rhIGF-1 continued on treatment for five years, when he elected to discontinue treatment after reviewing current growth trajectory and skeletal maturation. His untreated sibling was followed for four years through completion of growth.
Measure: Number; unit: standard deviation score
Arm/Group | Treatment With rhIGF-1 | Untreated Comparison
Number analyzed (Participants) | 1 | 1
standard deviation score
  Baseline | -2.86 | -2.92
  Year 1 | -2.53 | -2.99
  Year 2 | -2.54 | -2.84
  Year 3 | -2.61 | -2.69
  Year 4 | -2.43 | -2.63
  Year 5: number analyzed (Participants) | 1 | 0
  Year 5 | -2.27 |

3. Secondary Outcome: Pharmacokinetic/Pharmacodynamic (PK/PD) Relationship
Description: Assess the PK/PD relationship (PD marker being IGFBP-3) annually while on treatment with rhIGF-1
Time Frame: Yearly until completion of the study, up to 6 years
Population: Biochemical measurements in patient treated with rhIGF-1 over five years.
Measure: Number; unit: ng/mL
Groups:
- Free IGF-I: free IGF-I levels in ng/mL
- IGF-I: Total IGF-I levels in ng/mL
- IGFBP-3: Total IGFBP-3 levels in ng/mL
- PAPP-A2: PAPP-A2 levels in ng/mL
Arm/Group | Free IGF-I | IGF-I | IGFBP-3 | PAPP-A2
Number analyzed (Participants) | 1 | 1 | 1 | 1
ng/mL
  Baseline | 0.79 | 546.8 | 10000 | 0.110
  Year 1 | 1.17 | 709.1 | 6362 | 0.190
  Year 2 | 4.03 | 814.4 | 4001 | 0.122
  Year 3 | 5.13 | 961.7 | 6953 | 0.077
  Year 4 | 6.75 | 1200 | 6956 | 0.050
  Year 5 | 16.80 | 1200 | 6053 | 0

4. Other Pre Specified Outcome: Glucose Pre- and Post-treatment With Recombinant Human IGF-I
Description: Observe nonparametric measures of glucose pre and post ongoing treatment with rhIGF-1. Oral glucose tolerance tests (OGTT) were performed annually during the five-year treatment period at pre-treatment (baseline) and post-initiation of treatment (after 12 months, 24 months, 36 months, 48 months, and 60 months).
Time Frame: Yearly until completion of the study, up to 6 years
Population: OGTT results at baseline, 12 months, 24 months, 36 months, 48 months, 60 months
Measure: Number; unit: mg/dL
Groups:
- OGTT - 0 Minutes: 0 minute glucose
- OGTT - 30 Minutes: 30 minute glucose
- OGTT - 60 Minutes: 60 minute glucose
- OGTT - 90 Minutes: 90 minute glucose
- OGTT - 120 Minutes: 120 minute glucose
Arm/Group | OGTT - 0 Minutes | OGTT - 30 Minutes | OGTT - 60 Minutes | OGTT - 90 Minutes | OGTT - 120 Minutes
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
mg/dL
  Baseline | 111.4 | 193.9 | 203.9 | 156.6 | 127.5
  12 Months | 84.1 | 144.1 | 78.8 | 96.9 | 90.6
  24 Months | 103.5 | 183.4 | 132.0 | 122.7 | 116.2
  36 Months | 103.9 | 185.6 | 153.8 | 126.0 | 104.3
  48 Months | 97.3 | 203.1 | 249.3 | 198.7 | 169.7
  60 Months | 93.1 | 198.9 | 224.5 | 199.3 | 151.6

5. Other Pre Specified Outcome: Insulin Metabolism Pre- and Post-treatment With Recombinant Human IGF-I
Description: Observe nonparametric measures of insulin metabolism in each individual pre (baseline) and post ongoing treatment with rhIGF-1. Oral glucose tolerance testing (OGTT) was performed pre-treatment (baseline) and post-treatment (after 12 months, 24 months, 36 months, 48 months, and 60 months).
Time Frame: Annually through completion of the study, up to 6 years
Population: insulin levels measured with OGTT
Measure: Number; unit: mcIU/mL
Groups:
- OGTT - 0 Minutes: 0 minute insulin
- OGTT - 30 Minutes: 30 minute insulin
- OGTT - 60 Minutes: 60 minute insulin
- OGTT - 90 Minutes: 90 minute insulin
- OGTT - 120 Minutes: 120 minute insulin
Arm/Group | OGTT - 0 Minutes | OGTT - 30 Minutes | OGTT - 60 Minutes | OGTT - 90 Minutes | OGTT - 120 Minutes
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
mcIU/mL
  Baseline | 18.3 | 88.1 | 113.2 | 131.9 | 107
  12 Months | 4.5 | 38.1 | 11.2 | 22.6 | 22.3
  24 Months | 8.7 | 51.2 | 33.8 | 26.9 | 25.8
  36 Months | 20.4 | 120.6 | 67.6 | 58.9 | 50.3
  48 Months | 12.3 | 102.3 | 116.3 | 114.1 | 134.4
  60 Months | 14.9 | 84.2 | 98.5 | 116.9 | 94.4

6. Other Pre Specified Outcome: Body Mass Index at Baseline and on Treatment With rhIGF-I
Description: Observe nonparametric measures of body composition pre (baseline) and post ongoing treatment with rhIGF-1 (assessed after 12 months, 24 months, 36 months, 48 months, and 60 months of rhIGF-1 treatment). BMI percentiles were determined utilizing Centers for Disease Control and Prevention growth charts.
Time Frame: Annually until completion of the study, up to 6 years
Measure: Number; unit: percentile
Groups:
- BMI Percentile: BMI percentile at baseline and while on treatment with rhIGF-1
Arm/Group | BMI Percentile
Number analyzed (Participants) | 1
percentile
  Baseline | 12.96
  Year 1 | 30.83
  Year 2 | 56.60
  Year 3 | 42.76
  Year 4 | 54.20
  Year 5 | 70.42

7. Other Pre Specified Outcome: Body Composition at Baseline and on Treatment With rhIGF-I
Description: Observe nonparametric measures of body composition pre (baseline) and post ongoing treatment with rhIGF-1 (assessed after 12 months, 24 months, 36 months, 48 months, and 60 months of rhIGF-1 treatment). Body fat content and lean body mass were evaluated with dual energy x-ray absorptiometry.
Time Frame: Annually until completion of the study, up to 6 years
Measure: Number; unit: g
Groups:
- Total Lean Body Mass; Total Fat Mass: Body composition measures at baseline and while on treatment with rhIGF-1
Arm/Group | Total Lean Body Mass | Total Fat Mass
Number analyzed (Participants) | 1 | 1
g
  Baseline | 15274 | 6543
  Year 1 | 18961 | 7390
  Year 2 | 21366 | 10501
  Year 3 | 23876 | 10084
  Year 4 | 29779 | 12060
  Year 5 | 36398 | 13998

8. Other Pre Specified Outcome: Total Body Fat Percentage at Baseline and on Treatment With rhIGF-I
Description: as for outcome 7
Time Frame: Annually until completion of the study, up to 6 years
Measure: Number; unit: percentage of total body fat
Groups:
- Total Body Fat Percentage: Total body fat percentage at baseline and while on treatment with rhIGF-1
Arm/Group | Total Body Fat Percentage
Number analyzed (Participants) | 1
percentage of total body fat
  Baseline | 29.0
  Year 1 | 27.1
  Year 2 | 32.0
  Year 3 | 28.7
  Year 4 | 28.0
  Year 5 | 27.0

9. Other Pre Specified Outcome: C-telopeptide and Osteocalcin Concentrations at Baseline (Pre-treatment) and While on rhIGF-1.
Description: Observe nonparametric measures of bone turnover pre-treatment (baseline) and post initiation of ongoing treatment (at 12 months, 24 months, 36 months, 48 months, and 60 months) while on rhIGF-1
Time Frame: Yearly until completion of the study, up to 6 years
Measure: Number; unit: ng/mL
Groups:
- C-telopeptide; Osteocalcin: Bone turnover markers at baseline and while on rhIGF-1 therapy
Arm/Group | C-telopeptide | Osteocalcin
Number analyzed (Participants) | 1 | 1
ng/mL
  Baseline | 1744 | 86
  Year 1 | 2262 | 123
  Year 2 | 1762 | 88
  Year 3 | 2098 | 110
  Year 4 | 3216 | 152
  Year 5 | 2729 | 126

10. Other Pre Specified Outcome: Bone Density Pre-treatment (Baseline) and on Treatment With rhIGF-1
Description: Observe nonparametric measures of bone density at baseline (pre-treatment) and post initiation of ongoing treatment with rhIGF-1. Dual energy x-ray absorptiometry (DXA) was performed of total body less head, lumbar spine, hip, and forearm. Results are reported as height adjusted z-scores for age and gender, commonly done for bone density. A z-score of 0 is equivalent to population mean, positive above the mean, and negative below the mean. Z-scores within 2 standard deviations of the mean (Z-score 2 to -2) are generally considered normal, however are not sufficient to comment on presence or absence of osteoporosis in the pediatric population.
Time Frame: Annually until completion of therapy, up to 6 years
Measure: Number; unit: z-score
Groups:
- DXA Total Body Less Head; DXA Lumbar Spine; DXA Hip; DXA Forearm: Dual energy x-ray absorptiometry (DXA) at baseline and annually during give years of rhIGF-1 treatment
Arm/Group | DXA Total Body Less Head | DXA Lumbar Spine | DXA Hip | DXA Forearm
Number analyzed (Participants) | 1 | 1 | 1 | 1
z-score
  Baseline | -0.9 | -0.2 | -0.6 | -0.6
  Year 1 | -0.2 | 0.3 | -0.5 | -0.1
  Year 2 | -0.2 | 0.7 | -0.4 | -0.4
  Year 3 | -0.3 | 0.5 | -0.3 | -1.0
  Year 4 | -0.5 | 0.4 | -0.7 | -1.0
  Year 5 | -0.9 | 0.2 | -0.9 | -0.8

11. Other Pre Specified Outcome: Pharmacokinetic Description After Receiving Recombinant Human Insulin Like Growth Factor 1 (rhIGF-1): Maximum Corrected Total IGF-I and Free IGF-I
Description: This was a pharmacokinetic assessment in regards to rhIGF-1 completed in siblings with PAPP-A2 deficiency, Participants received a 120 mcg/kg dose of rhIGF-1 (Increlex). Pharmacokinetic measurements were obtained over 24 hours. To isolate the effect of injected rhIGF-1, baseline-corrected concentrations were included by subtracting baseline concentration from measured concentrations. Results reported include maximum corrected total IGF-I and free IGF-I. Due to constraints of reporting platform, time to maximum values and area under the curve (AUC) 12 hours after the dose are reported as separate outcomes.
Time Frame: At baseline, prior to the ongoing treatment phase with rhIGF-1
Measure: Mean (Full Range); unit: mcg/L
Groups:
- Healthy Controls: Healthy controls between the ages of 18-30 will be included in the 24-hour pharmacokinetic study.
Arm/Group | PAPP-A2 Deficient Patients | PAPP-A2 Heterozygous Relatives | Healthy Controls
Number analyzed (Participants) | 3 | 2 | 2
mcg/L
  Maximum corrected total IGF-I | 225 [186 to 254] | 243 [203 to 283] | 284.5 [278 to 291]
  Maximum corrected free IGF-I | 32 [26.6 to 35] | 30.5 [28.6 to 32.4] | 33.5 [10.9 to 56]

12. Other Pre Specified Outcome: Pharmacokinetic Description After Receiving Recombinant Human Insulin Like Growth Factor 1 (rhIGF-1): Time to Maximum Corrected Total IGF-I and Free IGF-I
Description: This was a pharmacokinetic assessment in regards to rhIGF-1 completed in siblings with PAPP-A2 deficiency, Participants received a 120 mcg/kg dose of rhIGF-1 (Increlex). Pharmacokinetic measurements were obtained over 24 hours. To isolate the effect of injected rhIGF-1, baseline-corrected concentrations were included by subtracting baseline concentration from measured concentrations. Results reported include time to maximum corrected total IGF-I and free IGF-I. Due to constraints of reporting platform, maximum corrected total IGF-I and free IGF-I values and area under the curve (AUC) 12 hours after the dose are reported as separate outcomes.
Time Frame: At baseline, prior to the ongoing treatment phase with rhIGF-1
Measure: Mean (Full Range); unit: h
Arm/Group | PAPP-A2 Deficient Patients | PAPP-A2 Heterozygous Relatives | Healthy Controls
Number analyzed (Participants) | 3 | 2 | 2
h
  Time to maximum corrected total IGF-I | 4.2 [3.5 to 5] | 3.3 [3 to 3.5] | 5.5 [5 to 6]
  Time to maximum corrected free IGF-I | 2.0 [1 to 3.5] | 2.3 [2 to 2.5] | 2.3 [2 to 2.5]

13. Other Pre Specified Outcome: Pharmacokinetic Description After Receiving Recombinant Human Insulin Like Growth Factor 1 (rhIGF-1): Area Under the Curve
Description: This was a pharmacokinetic assessment in regards to rhIGF-1 completed in siblings with PAPP-A2 deficiency, Participants received a 120 mcg/kg dose of rhIGF-1 (Increlex). Pharmacokinetic measurements were obtained over 24 hours. To isolate the effect of injected rhIGF-1, baseline-corrected concentrations were included by subtracting baseline concentration from measured concentrations. Results reported include area under the curve (AUC) 12 hours after the dose. Due to constraints of reporting platform, maximum corrected total IGF-I and free IGF-I, as well as time to maximum values separate outcomes.
Time Frame: At baseline, prior to the ongoing treatment phase with rhIGF-1
Measure: Mean (Full Range); unit: mcg*h/L
Arm/Group | PAPP-A2 Deficient Patients | PAPP-A2 Heterozygous Relatives | Healthy Controls
Number analyzed (Participants) | 3 | 2 | 2
mcg*h/L
  AUC_total IGF-1_0-12h | 2118 [1602 to 2406] | 2405 [2068 to 2742] | 2878.5 [2755 to 3002]
  AUC_free IGF-I_0-12h | 115.7 [95 to 133] | 135 [118 to 152] | 155.5 [64 to 247]

ADVERSE EVENTS:
Time Frame: The study adverse event data was collected over a period of 6 years (from baseline visit to one year post-treatment phone follow up).
Groups:
- Healthy Control Participants: Healthy controls between the ages of 18-30.
Arm/Group | PAPP-A2 Deficient Patients | PAPP-A2 Heterozygous Relatives | Healthy Control Participants
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 0/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAPP-A2 Deficient Patients (N=3) | PAPP-A2 Heterozygous Relatives (N=2) | Healthy Control Participants (N=2)
Pseudotumor cerebri in subject (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAPP-A2 Deficient Patients (N=3) | PAPP-A2 Heterozygous Relatives (N=2) | Healthy Control Participants (N=2)
Walking pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headaches (Nervous system disorders) | 1 (6) | 0 (0) | 0 (0)
Hair loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (Infections and infestations) | 1 (9) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (10) | 0 (0) | 0 (0)
Body aches and chills (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mild lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flu type A (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Viral strep throat (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Leg pain with walking (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Thrush on tongue (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Otitis externia (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Priaprism (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT02636270/Prot_SAP_002.pdf
  • Informed Consent Form (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT02636270/ICF_001.pdf